CLINICAL TRIAL: NCT04373915
Title: Improving Family Engagement With Remote Rounding in the NICU
Brief Title: Evaluating Parent Engagement, Attachment, Stress, and Satisfaction With Remote Rounding in the NICU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low participation in intervention
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Carly Dykstra, Neonatology Fellow, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY20181178
Record Dates: First submitted 2019-04-18; First posted 2020-05-05 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Parent Engagement; Parent Attachment; Parent Stress
Keywords: NICU; parent engagement; parent attachment; parent stress; remote rounding; video rounding

STUDY DESIGN:
Intervention Model Description: This is a single site prospective cohort study. Participants will be block randomized to standard rounding or availability of remote rounding based on their medical care team in the NICU. Parents using remote rounding will be compared to those who do not utilize remote rounding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Bedside Rounding (No Intervention)
- Remote Bedside Rounding (Experimental): Parents of infants on one care team will have the opportunity to participate in rounds via secure remote video software.
  Interventions: Behavioral: Remote Bedside Rounding

INTERVENTIONS:
Behavioral: Remote Bedside Rounding — Parents of infants on the medical team utilizing remote rounding will have the opportunity to participate in rounds by video conferencing at the infant's bedside. Participation will be tracked and surveys regarding stress, satisfaction, and attachment will be completed by parents in both groups.
  Arms: Remote Bedside Rounding

SUMMARY:
The admission of a newborn child to the neonatal intensive care unit (NICU) is among the most distressing situations that parents can face. There are many sources of parental stress including loss of control and competing demands outside of the NICU involving work and other children. During a prolonged admission it is often difficult for families to be present at bedside rounds on a daily basis and thus more difficult to discuss and collaborate with families in the care of their child. Healthcare has been slower than many other fields to adapt to the availability of new technology. This study hypothesizes that the use of wireless technology to allow parents to remotely participate on rounds would improve parental stress and satisfaction, in addition to improving engagement and attachment to their infant.

DETAILED DESCRIPTION:
Every year 10 to 15 percent of infants born in the United States, totaling roughly half a million babies, are admitted to a Neonatal Intensive Care Unit (NICU). Although survival rates are generally high, as many as half of these infants require a prolonged hospital stay. For parents, the admission of a newborn to the NICU is among the most emotionally distressing situations that they can face. A prolonged hospital stay can further impact the mother and family physically, psychologically, and financially.

During admission in the NICU it is often difficult for families to be present at bedside rounds on a daily basis due to transportation challenges or competing demands of work and care for siblings. Conflicting schedules between families and doctors make it more difficult to discuss and collaborate with families in the care of their child. The investigators hypothesize that this deficiency of communication and perceived loss of control can have significant impacts on maternal stress, satisfaction, engagement, and attachment.

Outside of the medical field, technology continues to advance as rapidly as ever. The medical field continues to struggle with adapting and using new technology and continue to lag behind many other fields. In recent years telemedicine has been used to facilitate patient care delivery, improve accessibility of health care services, and reduce healthcare costs however this use remains largely in the outpatient sector.

In the Neonatal Intensive Care Unit, Telemedicine has been used by one group to improve parent satisfaction in a variety of areas. A pilot study of the concept of remote or virtual rounding in a Pediatric Intensive Care Unit has been recently published in the literature. This project seeks to expand upon this knowledge to define and measure the impact on several aspects of neonatal care.

ELIGIBILITY:
Inclusion Criteria:

1. Parents with an infant admitted to the NICU/R4 with an anticipated length of stay of 2 weeks or more
2. Parent consents to study and answering questionnaires
3. English speaking
4. Infant is assigned to red or purple medical service team.
5. Infant age at enrollment: zero to 14 days old

Exclusion Criteria:

1. Parents with an infant admitted to the NICU/R4 with an anticipated length of stay less than 2 weeks
2. Parent is not willing to answer questionnaires
3. Non-English speaking
4. Patient is not assigned to red or purple medical service team.
5. Discharge to other than biological parents expected

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Parent Engagement | up to 1 year.
  Calendars will be placed at each infant's bedside to record engagement events consisting of participation in rounds, phone calls, visits, and kangaroo care. Each parental interaction recorded on the calendar will be counted. The mean and standard deviation of interactions over the study period will be calculated for each arm.

SECONDARY OUTCOMES:
Parent Satisfaction: survey | up to 6-10 weeks
  A short investigator created satisfaction survey will be used to measure parent satisfaction. Each question on the parent satisfaction survey will be analyzed separately and compared between the two groups. A Mann-Whitney U test will be used for each of the 8 likert questions.
Parent Stress | up to 6-10 weeks
  The Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU) will be used to measure parent stress. The instrument is a 46-item scale with 3 sub scales: infant behavior and appearance, parental role alteration, and sights and sounds. Each item is scored 1-5 on a likert scale (total sore range 46-230) with higher scores relating to higher stress. A standard t-test will be used.
Parent Attachment survey | up to 6-10 weeks
  The Maternal Attachment Inventory will be used to measure parent-infant attachment. This is a 26 item scale with each item scoring 1-4, for a total possible score of 26-104 with a higher score showing better attachment. Differences in attachment between the two arms will be assessed using a Wilcoxon rank sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Kuper-Sasse, MD, Principal Investigator — Rainbow Babies and Children's Hospital
Locations (1):
- Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miles MS, Funk SG, Carlson J. Parental Stressor Scale: neonatal intensive care unit. Nurs Res. 1993 May-Jun;42(3):148-52. PMID 8506163
- [Background] Muller ME. A questionnaire to measure mother-to-infant attachment. J Nurs Meas. 1994 Winter;2(2):129-41. PMID 7780768
- [Background] Gray JE, Safran C, Davis RB, Pompilio-Weitzner G, Stewart JE, Zaccagnini L, Pursley D. Baby CareLink: using the internet and telemedicine to improve care for high-risk infants. Pediatrics. 2000 Dec;106(6):1318-24. doi: 10.1542/peds.106.6.1318. PMID 11099583
- [Background] Epstein EG, Sherman J, Blackman A, Sinkin RA. Testing the Feasibility of Skype and FaceTime Updates With Parents in the Neonatal Intensive Care Unit. Am J Crit Care. 2015 Jul;24(4):290-6. doi: 10.4037/ajcc2015828. PMID 26134328
- [Background] Yager PH, Clark M, Cummings BM, Noviski N. Parent Participation in Pediatric Intensive Care Unit Rounds via Telemedicine: Feasibility and Impact. J Pediatr. 2017 Jun;185:181-186.e3. doi: 10.1016/j.jpeds.2017.02.054. Epub 2017 Mar 28. PMID 28363361